CLINICAL TRIAL: NCT02830087
Title: The Effect of Tourniquet Time and Pressure on Intraoperative and Postoperative Performance, Function, Pain, and Complications in Primary Total Knee Arthroplasty.
Brief Title: Tourniquet Pressure in Primary Total Knee Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No patient follow-up
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00038367
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Tourniquets; Knee Arthroplasty, Total; Knee Replacement, Total
Keywords: randomized controlled trial; tourniquet; tourniquet cuff pressure; total knee arthroplasty; total knee replacement; pain, postoperative; range of motion, articular; blood loss, surgical; muscle strength, quadriceps; walking; manipulation, orthopedic/therapeutic use; wound healing/surgery
MeSH Terms: conditions — Pain, Postoperative; Blood Loss, Surgical

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (6):
- 220 mmHg tourniquet cuff pressure (Active Comparator): Thigh tourniquet cuff inflated to 220 mmHg.
  Interventions: Procedure: Tourniquet Cuff Pressure
- 250 mmHg tourniquet cuff pressure (Active Comparator): Thigh tourniquet cuff inflated to 250 mmHg
  Interventions: Procedure: Tourniquet Cuff Pressure
- 275 mmHg tourniquet cuff pressure (Active Comparator): Thigh tourniquet cuff inflated to 275 mmHg
  Interventions: Procedure: Tourniquet Cuff Pressure
- 300 mmHg tourniquet cuff pressure (Active Comparator): Thigh tourniquet cuff inflated to 300 mmHg
  Interventions: Procedure: Tourniquet Cuff Pressure
- 325 mmHg tourniquet cuff pressure (Active Comparator): Thigh tourniquet cuff inflated to 325 mmHg
  Interventions: Procedure: Tourniquet Cuff Pressure
- 350 mmHg tourniquet cuff pressure (Active Comparator): Thigh tourniquet cuff inflated to 350 mmHg
  Interventions: Procedure: Tourniquet Cuff Pressure

INTERVENTIONS:
Procedure: Tourniquet Cuff Pressure — Tourniquet cuff pressure is how hard the tourniquet cuff, which is placed around the patient's thigh, presses on the thigh in order to cut off blood supply to the lower leg during total knee surgery.

SUMMARY:
This proposed novel randomized control trial (RCT) seeks to address this gap in TKA protocol by gaining a better understanding of the relationship between tourniquet pressure and time, and intraoperative performance and post-operative outcomes. This study does not seek to answer the question of "tourniquet vs no tourniquet", but to seek a tourniquet usage that would maximize the intraoperative benefits for the surgeon and minimize the negative consequences for patient outcomes.

Specific Aim #1: enroll around 146 primary TKA patients.

Specific Aim #2: evaluate different tourniquet cuff pressures (TCP) and tourniquet times in relation to intraoperative performance.

Specific Aim #3: evaluate different TCP and tourniquet times in relation to post-operative pain and complications of short-term, intermediate, and long-term followup.

Specific Aim #4: evaluate different TCP and tourniquet times in relation to post-operative function of short-term, intermediate, and long-term followup.

DETAILED DESCRIPTION:
The overall goal of the project is to evaluate the relationship of two variables: 1) tourniquet cuff pressure (TCP); and 2) tourniquet time (i.e. duration of inflation) during primary TKA relative to three categories of outcomes: 1) intraoperative performance; 2) post-operative pain and complications; and 3) post-operative complications.

Design

This study will use a randomized controlled trial that is double-blinded. The co-investigator, Mark Nazal, along with the principal investigator, Dr. Maxwell Langfitt, will work with the Orthopaedic Clinic Research Coordinator to recruit around 146 patients. Mark Nazal will then randomize these patients into one of six tourniquet cuff pressure (TCP) groups:

1. 220 mmHg 4) 300 mmHg
2. 250 mmHg 5) 325 mmHg
3. 275 mmHg 6) 350 mmHg

The primary TKA procedure will be performed by one of the three fellowship-trained orthopedic surgeons at Wake Forest Baptist Hospital (Dr. Maxwell Langfitt, Dr. Jason Lang, and Dr. John Shields). The orthopedic surgeon and the patient will be blinded to the TCP assignment and will not be told what tourniquet pressure is being applied. The OR nursing team will be told what the patient's assigned TCP is in order to perform the actual inflation.

Data collection will include short-term data: post-operative day 1 (POD1), post-operative day 2 (POD2), and 2-week followup; intermediate data: 6-week and 12-week followup; and long-term data: 1-year followup.

The data collection for the first category of outcomes, intraoperative performance, will begin preoperatively, with the recording of baseline characteristics: circumference of the thigh in centimeters, baseline hemoglobin levels, and thromboembolism risk evaluation.

Intraoperative data will include: the type of anesthesia, the tourniquet size in centimeters, and whether or not a drain is inserted into the joint. The time of inflation and time of deflation will be noted in order to determine the duration of tourniquet inflation.

Then preincisional blood pressure (BP) will be measured and will continue to be noted every 15 minutes. At the conclusion of the procedure the surgeon will rate intraoperative bloodlessness on a four-point scale: 1-bloodless, 2-nearly bloodless, some bleeding; 3-bloody, tourniquet is no better than not using; or 4-venous tourniquet, tourniquet is making the procedure more difficult. Intraoperative bloodlessness is being used to determine the functionality and effectiveness of the tourniquet, surgical field visualization, and surgical site dryness.

The data collection for the second category of outcomes, post-operative pain and complications, will begin on post-operative day 1 (POD1). Post-operative (post-op) pain will be assessed using a 0-10 pain rating visual analog scale for both the knee and the thigh, and will be measured at POD1, POD2, 2-week followup, 6-week followup, 12-week followup, and 1-year followup. Next, wound healing issues will be assessed at POD1, POD2, 2-week followup, 6-week followup, and 12-week followup. Wound healing issues include blisters, wound drainage, thigh bruising, significant erythema, decreased peripheral pulse, evidence of decreased distal perfusion, or decreased distal sensation.13 Estimated total blood loss will be assessed at POD2 using pre-operative Hgb-level compared to Hgb-level on post-op day 2. The patient's estimated blood volume (EBV) will be calculated using Nadler's formulas for men and women.16

Then Meunier's formula will be used to calculate estimated blood loss.16 If a drain was inserted, then the volume of drainage will be measured at POD1. Finally, aseptic loosing of the implant leading to the need for revision will be assessed at 1-year followup.

The data collection for the third category of outcomes, post-operative function, will begin at POD1. Ability to ambulate will be measured in distance by feet at POD1 and POD2. Furthermore, assessment of any use of assisted device for ambulation (wheelchair, walker, 4-point cane, and 1-point cane) will be done at POD1, POD2, 2-week followup, 6-week followup, 12-week followup and 1-year followup. Quadriceps strength and range of motion (ROM) will be recorded at 2-week followup, 6-week followup, and 12-week followup. Quadriceps strength will be measured on a 5-point scale, where 0 is no movement and 5 is full strength. ROM will be measured in degrees of motion. Next, the necessity of performing a manipulation under anesthesia (MUA) due to limited joint motion will be recorded at 6-week followup and 12-week followup. The type of PT will be recorded at 2-week followup, 6-week followup, and 12-week followup. Types of PT include out-patient PT, home health PT, PT rehabilitation, and skilled nursing facility PT.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 80 years old
2. primary TKA, not revision

Exclusion Criteria:

1. systolic blood pressure (BP) ≥ 170 mmHg
2. one-staged bilateral TKA or stages less than three months apart
3. history of peripheral vascular disease
4. history of thromboembolism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09-20 (Actual); Study Completion 2016-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Holden, Study Director — Manager; Maxwell K Langfitt, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Davie Medical Center, Bermuda Run, North Carolina
  - Wake Forest Baptist Hospital, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang FZ, Zhong HM, Hong YC, Zhao GF. Use of a tourniquet in total knee arthroplasty: a systematic review and meta-analysis of randomized controlled trials. J Orthop Sci. 2015 Jan;20(1):110-23. doi: 10.1007/s00776-014-0664-6. Epub 2014 Nov 6. PMID 25373840
- [Background] Alcelik I, Pollock RD, Sukeik M, Bettany-Saltikov J, Armstrong PM, Fismer P. A comparison of outcomes with and without a tourniquet in total knee arthroplasty: a systematic review and meta-analysis of randomized controlled trials. J Arthroplasty. 2012 Mar;27(3):331-40. doi: 10.1016/j.arth.2011.04.046. Epub 2011 Sep 22. PMID 21944371
- [Background] Berry DJ, Bozic KJ. Current practice patterns in primary hip and knee arthroplasty among members of the American Association of Hip and Knee Surgeons. J Arthroplasty. 2010 Sep;25(6 Suppl):2-4. doi: 10.1016/j.arth.2010.04.033. Epub 2010 Jul 1. PMID 20580196
- [Background] Tai TW, Lin CJ, Jou IM, Chang CW, Lai KA, Yang CY. Tourniquet use in total knee arthroplasty: a meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2011 Jul;19(7):1121-30. doi: 10.1007/s00167-010-1342-7. Epub 2010 Dec 15. PMID 21161177
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Ledin H, Aspenberg P, Good L. Tourniquet use in total knee replacement does not improve fixation, but appears to reduce final range of motion. Acta Orthop. 2012 Oct;83(5):499-503. doi: 10.3109/17453674.2012.727078. Epub 2012 Sep 14. PMID 22974220
- [Background] Li B, Wen Y, Wu H, Qian Q, Lin X, Zhao H. The effect of tourniquet use on hidden blood loss in total knee arthroplasty. Int Orthop. 2009 Oct;33(5):1263-8. doi: 10.1007/s00264-008-0647-3. Epub 2008 Aug 27. PMID 18751703
- [Background] Liu D, Graham D, Gillies K, Gillies RM. Effects of tourniquet use on quadriceps function and pain in total knee arthroplasty. Knee Surg Relat Res. 2014 Dec;26(4):207-13. doi: 10.5792/ksrr.2014.26.4.207. Epub 2014 Dec 2. PMID 25505702
- [Background] Zhang W, Li N, Chen S, Tan Y, Al-Aidaros M, Chen L. The effects of a tourniquet used in total knee arthroplasty: a meta-analysis. J Orthop Surg Res. 2014 Mar 6;9(1):13. doi: 10.1186/1749-799X-9-13. PMID 24602486
- [Background] Ejaz A, Laursen AC, Kappel A, Laursen MB, Jakobsen T, Rasmussen S, Nielsen PT. Faster recovery without the use of a tourniquet in total knee arthroplasty. Acta Orthop. 2014 Aug;85(4):422-6. doi: 10.3109/17453674.2014.931197. Epub 2014 Jun 23. PMID 24954487
- [Background] Olivecrona C, Ponzer S, Hamberg P, Blomfeldt R. Lower tourniquet cuff pressure reduces postoperative wound complications after total knee arthroplasty: a randomized controlled study of 164 patients. J Bone Joint Surg Am. 2012 Dec 19;94(24):2216-21. doi: 10.2106/JBJS.K.01492. PMID 23318611
- [Background] Reilly CW, McEwen JA, Leveille L, Perdios A, Mulpuri K. Minimizing tourniquet pressure in pediatric anterior cruciate ligament reconstructive surgery: a blinded, prospective randomized controlled trial. J Pediatr Orthop. 2009 Apr-May;29(3):275-80. doi: 10.1097/BPO.0b013e31819bcd14. PMID 19305279
- [Background] Clarke MT, Longstaff L, Edwards D, Rushton N. Tourniquet-induced wound hypoxia after total knee replacement. J Bone Joint Surg Br. 2001 Jan;83(1):40-4. doi: 10.1302/0301-620x.83b1.10795. PMID 11245536
- [Background] Gibon E, Courpied JP, Hamadouche M. Total joint replacement and blood loss: what is the best equation? Int Orthop. 2013 Apr;37(4):735-9. doi: 10.1007/s00264-013-1801-0. Epub 2013 Feb 6. PMID 23385607
- See also: Citation #1 — https://www.uptodate.com/contents/total-knee-replacement-arthroplasty-beyond-the-basics?source=see_link
- See also: Citation #6 — https://www.hcup-us.ahrq.gov/reports/statbriefs/sb186-Operating-Room-Procedures-United-States-2012.jsp

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 220 mmHg Tourniquet Cuff Pressure | 250 mmHg Tourniquet Cuff Pressure | 275 mmHg Tourniquet Cuff Pressure | 300 mmHg Tourniquet Cuff Pressure | 325 mmHg Tourniquet Cuff Pressure | 350 mmHg Tourniquet Cuff Pressure
Started | 4 | 4 | 4 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 4 | 3 | 3 | 3
Not completed — No study staff to follow-up patients | 4 | 4 | 4 | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 220 mmHg Tourniquet Cuff Pressure | 250 mmHg Tourniquet Cuff Pressure | 275 mmHg Tourniquet Cuff Pressure | 300 mmHg Tourniquet Cuff Pressure | 325 mmHg Tourniquet Cuff Pressure | 350 mmHg Tourniquet Cuff Pressure | Total
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 3 | 2 | 3 | 0 | 14
  >=65 years | 2 | 0 | 1 | 1 | 0 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (6.7) | 58.3 (8.9) | 59.5 (8.9) | 63.7 (13.2) | 50.7 (7.2) | 73.7 (2.1) | 61.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 2 | 1 | 2 | 11
  Male | 1 | 3 | 2 | 1 | 2 | 1 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 4 | 3 | 3 | 3 | 21

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain
Description: Pain on a 11-point pain scale (0-10), with higher scores denoting worse outcomes
Time Frame: Postoperative Day 1 through two weeks
Population: data not collected for all participants
Measure: Number; unit: score on a scale
Arm/Group | 220 mmHg Tourniquet Cuff Pressure | 250 mmHg Tourniquet Cuff Pressure | 275 mmHg Tourniquet Cuff Pressure | 300 mmHg Tourniquet Cuff Pressure | 325 mmHg Tourniquet Cuff Pressure | 350 mmHg Tourniquet Cuff Pressure
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 1
score on a scale |  |  | 3 | 7 |  | 9

2. Secondary Outcome: Estimated Blood Loss
Description: Meunier's formula will be used to calculate estimated blood loss, comparing preoperative blood draw to postoperative day 2 blood draw.
Time Frame: Postoperative Day 2
Population: No data collected
Arm/Group | 220 mmHg Tourniquet Cuff Pressure | 250 mmHg Tourniquet Cuff Pressure | 275 mmHg Tourniquet Cuff Pressure | 300 mmHg Tourniquet Cuff Pressure | 325 mmHg Tourniquet Cuff Pressure | 350 mmHg Tourniquet Cuff Pressure
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Range of Motion
Description: Measure degrees of knee flexion
Time Frame: 2-week follow-up
Population: data not collected for all participants
Measure: Number; unit: Degrees
Arm/Group | 220 mmHg Tourniquet Cuff Pressure | 250 mmHg Tourniquet Cuff Pressure | 275 mmHg Tourniquet Cuff Pressure | 300 mmHg Tourniquet Cuff Pressure | 325 mmHg Tourniquet Cuff Pressure | 350 mmHg Tourniquet Cuff Pressure
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0
Degrees |  |  | 78 | 15 |  |

4. Secondary Outcome: Intra-operative Bloodlessness
Description: four-point scale:
  * 1 = bloodless
  * 2 = nearly bloodless, some bleeding
  * 3 = bloody, tourniquet no better than not using
  * 4 = venous tourniquet, tourniquet making things worse
  Higher scores denotes worse outcome
Time Frame: Intraoperative
Population: data not collected for all participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 220 mmHg Tourniquet Cuff Pressure | 250 mmHg Tourniquet Cuff Pressure | 275 mmHg Tourniquet Cuff Pressure | 300 mmHg Tourniquet Cuff Pressure | 325 mmHg Tourniquet Cuff Pressure | 350 mmHg Tourniquet Cuff Pressure
Number analyzed (Participants) | 0 | 1 | 1 | 2 | 0 | 0
score on a scale |  | 1 (NA) — Standard Deviation is not calculable for 1 participant | 1 (NA) — Standard Deviation is not calculable for 1 participant | 2 (1.4) |  |

5. Secondary Outcome: Number of Participants With Wound Healing Issues
Description: Any wound issues including blisters, wound drainage, thigh bruising, significant erythema, decreased peripheral pulse, evidence of decreased distal perfusion, or decreased distal sensation
Time Frame: Postoperative Day 1 through 12 week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | 220 mmHg Tourniquet Cuff Pressure | 250 mmHg Tourniquet Cuff Pressure | 275 mmHg Tourniquet Cuff Pressure | 300 mmHg Tourniquet Cuff Pressure | 325 mmHg Tourniquet Cuff Pressure | 350 mmHg Tourniquet Cuff Pressure
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Need for Revision of Total Knee Arthroplasty
Description: Number of participants that needed a revision was necessary within one year
Time Frame: One Year Follow-up
Population: No data collected
Arm/Group | 220 mmHg Tourniquet Cuff Pressure | 250 mmHg Tourniquet Cuff Pressure | 275 mmHg Tourniquet Cuff Pressure | 300 mmHg Tourniquet Cuff Pressure | 325 mmHg Tourniquet Cuff Pressure | 350 mmHg Tourniquet Cuff Pressure
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Ability to Ambulate
Description: Distance Walked in Feet
Time Frame: Postoperative Day 1 through Postoperative Day 2
Population: data not collected for all participants
Measure: Number; unit: Feet
Arm/Group | 220 mmHg Tourniquet Cuff Pressure | 250 mmHg Tourniquet Cuff Pressure | 275 mmHg Tourniquet Cuff Pressure | 300 mmHg Tourniquet Cuff Pressure | 325 mmHg Tourniquet Cuff Pressure | 350 mmHg Tourniquet Cuff Pressure
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
Feet |  |  | 208 |  |  |

8. Secondary Outcome: Quadriceps Strength
Description: Six Point Strength Scale 0 - No muscle movement
  1. -Muscle movement, without movement at the joint
  2. -Movement at the joint, but not against gravity
  3. -Movement against gravity, but not against resistance
  4. -Movement against resistance, but less than full strength
  5. -Full Strength
  Higher scores denotes better outcome
Time Frame: 2-week follow-up through 12-week follow-up
Population: data not collected for all participants
Measure: Number; unit: score on a scale
Arm/Group | 220 mmHg Tourniquet Cuff Pressure | 250 mmHg Tourniquet Cuff Pressure | 275 mmHg Tourniquet Cuff Pressure | 300 mmHg Tourniquet Cuff Pressure | 325 mmHg Tourniquet Cuff Pressure | 350 mmHg Tourniquet Cuff Pressure
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
score on a scale |  |  | 4 |  |  |

9. Secondary Outcome: Need for Manipulation Under Anesthesia
Description: Number of participants that needed a manipulation under anesthesia was necessary within 12 weeks
Time Frame: 6-week follow-up through 12-week follow-up
Population: No data collected
Arm/Group | 220 mmHg Tourniquet Cuff Pressure | 250 mmHg Tourniquet Cuff Pressure | 275 mmHg Tourniquet Cuff Pressure | 300 mmHg Tourniquet Cuff Pressure | 325 mmHg Tourniquet Cuff Pressure | 350 mmHg Tourniquet Cuff Pressure
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 4 months
Arm/Group | 220 mmHg Tourniquet Cuff Pressure | 250 mmHg Tourniquet Cuff Pressure | 275 mmHg Tourniquet Cuff Pressure | 300 mmHg Tourniquet Cuff Pressure | 325 mmHg Tourniquet Cuff Pressure | 350 mmHg Tourniquet Cuff Pressure
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/3 | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
The trial had limited patient enrollment, randomization, and follow-up due to limited study staff.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No